CLINICAL TRIAL: NCT02531282
Title: Effect of and Experiences With a Health Promotion Intervention for People With Chronic Pain at a Healthy Life Centre - an Open, Pragmatic, Randomized Controlled Trial With a Nested Qualitative Study
Brief Title: Effect of a Health Promotion Intervention for People With Chronic Pain at a Healthy Life Centre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Trondheim Kommune (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015/1030
Record Dates: First submitted 2015-08-21; First posted 2015-08-24 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Chronic Pain
Keywords: Patient education as topic; Health promotion; Patient participation; Self efficacy
MeSH Terms: conditions — Chronic Pain; Patient Participation | interventions — Patient Education as Topic; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health promotion in patient education (Experimental): The self-management patient education has been developed at the Healthy Life Centre in Trondheim municipality based on cognitive behavioural theory and psychomotor physiotherapy. The intervention is developed in a health promotion framework focusing on salutogenesis aiming to improve the participants ability to activate their own resources for health behaviour changes .
  Interventions: Behavioral: Patient education
- Physical activity in groups (Active Comparator): Physical activity once a week for a period of 6 weeks in form of walking and simple strength exercises outdoor in groups led by an instructor. .
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Patient education — Self-management patient education in groups once a week for 6 weeks. Each session include pain-related theory, group discussions and physical exercises focusing on posture and relaxation. Instructors with education in health promotion and behavioural change in addition to psychomotor physiotherapy.
  Arms: Health promotion in patient education
Behavioral: Physical activity — Physical activity once a week for a period of 6 weeks in form of walking and simple strength exercises outdoor in groups led by an instructor. Each session has a duration of one hour. The instructor has education in physical activity.
  Arms: Physical activity in groups

SUMMARY:
The study's primary objective is to test the hypothesis that a group-based health promotion intervention with patient education and practical exercises delivered at a Healthy Life Centre increases patient activation in people living with chronic pain. Due to many people living with chronic pain, interventions focusing on self-management and coping are on the agenda in primary care. This study will investigate whether a Healthy Life Centre in a municipality is a suitable setting for interventions targeting people living with chronic pain. Short and long term effect of an intervention developed in a health promotion and salutogenic framework will be investigated in a randomized clinical trial.

DETAILED DESCRIPTION:
Previous research indicates that if self-management interventions are developed within a health promotion framework focusing on the participants' strengths, there is a beneficial effect on patient activation and thus on self-management behaviour. However, there is a lack of knowledge about which interventions will improve patient activation for persons with chronic pain. To be sustainable, such interventions should be delivered using the least possible amount of resources needed to get an effect. One way to do so is to deliver the intervention in primary care instead of in hospitals. The Healthy Life Centre is ideally situated to deliver these interventions. This is especially true due to their task of focusing on health promotion but also because they are set up to deliver low level interventions, meaning that it should be easy for everyone to access their services.

ELIGIBILITY:
Inclusion Criteria:

* pain for 3 months or more
* able to participate in one hour physical activity

Exclusion Criteria:

* not fluent in Norwegian
* chronic pain arising from active malignant disease
* serious mental health illness
* substance abuse issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM)- 13 items | 1 year
  Self-reported questionnaire at baseline, and 3- 6- 12 months after intervention. PAM-13 is an interval-level, uni-dimensional measure questionnaire with a four point scale with an additional not applicable option, giving a raw score from 13- 52, which is calibrated to a total score between 0 (less activated) to 100 (most activated).

SECONDARY OUTCOMES:
Sense of Coherence (SOC) according to SOC-13 questionnaire | 1 year
  Self-reported questionnaire, The SOC-13, at baseline, and 3-6-12 months after intervention. The questionnaire consists of 13 items with seven options for answers, each with a scoring range from 1 to 7, giving a total score from 13 to 91.
Psychological distress on the Hospital Anxiety and Depression Scale (HADS) | 1 year
  Self-reported questionnaire, the Hospital Anxiety and Depression Scale (HADS) at baseline, and 3-6-12 months after intervention. The questionnaire consists of 14 items producing a separate score for anxiety and depression. The instrument has a total range from 0 (best) to 42 (worst).
Pain severity in Brief Pain Questionnaire | 1 year
  Self-reported pain severity measured by 4 questions in the Brief Pain Inventory (BPI) instrument. All items in BPI are scored using a numeric rating scale from 0 to 10. Measured at baseline, and 3-6-12 months after intervention.
Pain interference in Brief Pain Questionnaire | 1 year
  Self-reported pain interference measured by 7 questions in the Brief Pain Inventory (BPI) instrument. All items in BPI are scored using a numeric rating scale from 0 to 10. Measured at baseline, and 3-6-12 months after intervention.
Pain intensity on a Visual Analogue Scale 100-mm | 1 year
  Self-reported experience of pain during the previous week using a one-item 100 mm Visual Analogue Scale at baseline, and 3-6-12 months after intervention. The anchoring points are "no pain" (0) and "intolerable pain" (100).
Quality of Life on EuroQoL (EQ-5D-5L) Instrument | 1 year
  Self-reported using the EQ-5 Dimensional instrument. Measured at baseline, and 3-6-12 months after intervention.
Well-being on Visual Analogue Self-Rating Scale 100-mm | 1 year
  Self-reported well-being measured by the Arizona Integrative Outcome Scale (AIOS) at baseline, and 3-6-12 months after intervention. This is a one-item 100 mm long Visual Analogue Self-Rating Scale followed by an instruction to reflect on the sense of well-being during the last month. The anchoring points are "worst you have ever been (0) and "best you ever been" (100).
Pain related self-efficacy according to Pain Self-efficacy Questionnaire (PSEQ) | 1 year
  Self-reported pain self-efficacy using the instrument Pain Self-efficacy Questionnaire (PSEQ) at baseline, and 3-6-12 months after intervention. The questionnaire consist of 10 items scored on a range from 0 to 60, with higher scores indicating stronger self-efficacy beliefs.
Physical ability in 30-seconds chair-to-stand test. | 1 year
  The 30 seconds chair to stand test (30CST) performed at baseline, and 3-6-12 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Grønning, phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- Trondheim Kommune, Friskliv og mestring, Trondheim, Norway

REFERENCES:
- [Background] Nost TH, Steinsbekk A, Bratas O, Gronning K. Expectations, effect and experiences of an easily accessible self-management intervention for people with chronic pain: study protocol for a randomised controlled trial with embedded qualitative study. Trials. 2016 Jul 18;17(1):325. doi: 10.1186/s13063-016-1462-6. PMID 27430319
- [Result] Nost TH, Steinsbekk A, Bratas O, Gronning K. Short-term effect of a chronic pain self-management intervention delivered by an easily accessible primary healthcare service: a randomised controlled trial. BMJ Open. 2018 Dec 9;8(12):e023017. doi: 10.1136/bmjopen-2018-023017. PMID 30530580
- [Result] Nost TH, Steinsbekk A, Bratas O, Gronning K. Twelve-month effect of chronic pain self-management intervention delivered in an easily accessible primary healthcare service - a randomised controlled trial. BMC Health Serv Res. 2018 Dec 29;18(1):1012. doi: 10.1186/s12913-018-3843-x. PMID 30594190
- [Derived] Nost TH, Steinsbekk A, Riseth L, Bratas O, Gronning K. Expectations towards participation in easily accessible pain management interventions: a qualitative study. BMC Health Serv Res. 2017 Nov 10;17(1):712. doi: 10.1186/s12913-017-2668-3. PMID 29126444